CLINICAL TRIAL: NCT05554965
Title: Clinical Study of Remazolam Besylate for Sedation During Endoscopic Hemostatic Treatment of Esophageal and Gastric Variceal Bleeding
Brief Title: Endoscopic Hemostatic and Sedative Treatment of Esophageal and Gastric Variceal Bleeding
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20220819
Record Dates: First submitted 2022-09-15; First posted 2022-09-26 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-08

CONDITIONS: Endoscopic Hemostasis; Sedation
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol (Active Comparator): The control group was sedated with propofol
  Interventions: Drug: Propofol
- Remimazolam besylate (Experimental): The experimental group was given remazolam besylate for sedation
  Interventions: Drug: Remimazolam besylate

INTERVENTIONS:
Drug: Propofol — Remifentanil maintenance analgesic dose was 1.2-9 μg/kg/h. If the CPOT score ≥3 at the time of maintenance administration, dose adjustment can be considered. Propofol was used for sedation at a loading dose of 0.5mg/kg and a maintenance dose of 1.5mg/kg/h.
  Other Names: Active Comparator
  Arms: propofol
Drug: Remimazolam besylate — Remifentanil was administered at a maintenance dose of 1.2-9 μg/kg/h for analgesia. If CPOT score ≥3 during maintenance administration, dose adjustment could be considered. For sedation, remazolam besylate was given a load of 0.1-0.2mg/kg and a maintenance dose of 0.1-0.3mg/kg/h.
  Other Names: Experimental
  Arms: Remimazolam besylate

SUMMARY:
Remazolam besylate was used for sedation during endoscopic hemostasis in patients with esophageal and gastric varices rupture and bleeding in liver cirrhosis. The onset time, recovery time and incidence of adverse reactions were observed.

DETAILED DESCRIPTION:
Esophagogastric variceal bleeding (EGVB) is one of the most serious and common complications of liver cirrhosis. Endoscopic hemostasis is the most widely used and important method for the prevention and treatment of EGVB. The treatment of varicose veins hemostasis under gastroscope has the problem of long operation time. Patients are prone to nausea, vomiting and excessive secretions due to nervousness and fear, which affect endoscopic insertion and observation, leading to failure of ligation and massive bleeding, and even death. Therefore, appropriate analgesic and sedative drugs are necessary to ensure endoscopic treatment and improve the prognosis. Remimazolam, an ultra-short-acting benzodiazepine drug, is obtained by introducing metabolizable methyl propionate side chain into midazolam. It may have a good effect on sedation during endoscopic hemostasis in cirrhotic patients with ruptured esophageal and gastric varices.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with bleeding from ruptured esophageal and gastric varices
* Endoscopic hemostatic treatment was performed
* Body Mass Index(BMI)18～28kg/m2

Exclusion Criteria:

* History or evidence of increased risk of sedation/anesthesia;
* Pregnant and lactating women;
* Have participated in other drug trials within 30 days prior to enrollment;
* those with contraindications to propofol, opioids and their remedies;
* Unwilling to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Sedation scores | From the begin to 48 hours after procedure
  sedation scores were performed during administration,Richmond Agitation-Sedation Scale（RASS）1~-2 was defined as compliance,Otherwise, sedation was considered inadequate

SECONDARY OUTCOMES:
Rate of adverse events | Within 2 hours from the start of administration to the end of administration
  Any adverse events that occurred during the administration of the drug, such as bradycardia, hypotension, respiratory depression, etc
Vital signs | From the begin to 48 hours after procedure
  Systolic and Diastolic Blood Pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared with team members
Supporting Information: Study Protocol, SAP, ICF, CSR